CLINICAL TRIAL: NCT03509987
Title: The Evaluation of Point of Care Testing for Determining Hemoglobin Levels in Geriatric Intensive Care Patients
Acronym: hb levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, MEHTAP HONCA, MD, Director, Kecioren Education and Training Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KeciorenTRH
Record Dates: First submitted 2018-04-16; First posted 2018-04-27 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Point-of-Care Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- hb analysis with Hemacue (Other): Hb analysis with Hemacue and with arterial blood gas analyser in geriatric ill patients requiring intensive care
  Interventions: Device: HemaCue

INTERVENTIONS:
Device: HemaCue — comparing hemoglobin (Hb) levels determined by point of care testing HemaCue and arterial blood gas analyzer with an automated hematology analyzer in critically ill geriatric patients.
  Other Names: Blood gas analyser

SUMMARY:
The aim of the present study was to compare hemoglobin (Hb) levels determined by point of care testing HemaCue and arterial blood gas analyzer with an automated hematology analyzer in critically ill geriatric patients.Forty geriatric patients requiring intensive care treatment were included in the study. Arterial blood sample was analyzed using HemaCue (HbHemaCueArterial), blood gas analyzer (Techno Medica, Gastat1800 series) (HbBGA) and an automated hematology analyzer (Cell Dyne 3700 System, Abbot Laboratories)(HbLab) as a reference method. Capillary blood measurements were performed (HbHemaCueCapillary) by HemaCue at bedside.

DETAILED DESCRIPTION:
The aim of the present study was to compare hemoglobin (Hb) levels determined by point of care testing HemaCue and arterial blood gas analyzer with an automated hematology analyzer in critically ill geriatric patients.Forty geriatric patients requiring intensive care treatment were included in the study. Arterial blood sample was analyzed using HemaCue (HbHemaCueArterial), blood gas analyzer (Techno Medica, Gastat1800 series) (HbBGA) and an automated hematology analyzer (Cell Dyne 3700 System, Abbot Laboratories)(HbLab) as a reference method. Capillary blood measurements were performed (HbHemaCueCapillary) by HemaCue at bedside. Bland Altman Analysis was applied to the results .

ELIGIBILITY:
Inclusion Criteria:

* geriatric patients requiring intensive care treatment

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
hemoglobin levels | 1 months
  comparing hemoglobin (Hb) levels determined by point of care testing HemaCue and arterial blood gas analyzer with an automated hematology analyzer in critically ill geriatric patients.

CONTACTS AND LOCATIONS:
Overall Officials: MEHTAP HONCA, Ass. Prof, Principal Investigator — Kecioren training and research Hospital , Department of Anesthesiology and Reanimation
Locations (1):
- Mehtap Honca, Ankara, Kecioren, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No